CLINICAL TRIAL: NCT04070066
Title: Educational Strategy for the Development of Skills in Exchange Trnasfusion: a Randomized Clinical Trial Protocol
Brief Title: Educational Strategy in Exchange Transfusion
Acronym: INTEXUS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de la Sabana (Other)
Responsible Party: Principal Investigator, sergio Ivan agudelo Perez, Professor, Universidad de la Sabana
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 451
Record Dates: First submitted 2019-08-22; First posted 2019-08-28 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2025-01

CONDITIONS: Newborn Morbidity; Simulation Training; Telemedicine; Assessment, Self
Keywords: Newborn, infant; exchange-transfusion

STUDY DESIGN:
Intervention Model Description: For the assignment of the students to the study groups, a randomization sequence will be generated through a computer-generated process. This process will be centralized in the paediatric office of the Universidad de La Sabana (University of La Sabana). The sequence will be generated through the Research Randomizer page (www.randomizer.org), and a permuted blocks strategy with block size of eight (8) will be used. The permuted blocks strategy and the size of the blocks will not be known by the researcher. To ensure the concealment of the random sequence, it will be placed in opaque envelopes at the time of assignment.
Who Masked: Outcomes Assessor
Masking Description: Due to the nature of the interventions, masking cannot be applied to the researcher or the student. However, blinding will be applied to the research team responsible for data analysis and to the expert neonatologist who will perform the evaluations of the video recorded procedures using the checklist. The database will be coded, and the identification code will not be available to the analyst.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Digital didactic environment (Experimental): Students assigned to this group will receive access to a digital didactic environment where they will have at their disposal the exchange transfusion guide and a complete video explaining the indications, the preparation of supplies and the newborn for the procedure, the management of medical devices required and a step-by-step description of the exchange transfusion technique. Finally, the student will see an integrated clinical case. This video will be developed by the neonatology and paediatric medical education teaching team in the simulation laboratory of the university using neonatal high-fidelity simulators, a simulated mother and the necessary medical equipment and supplies.
  Interventions: Other: Digital didactic environment
- • Simulated scenario (Active Comparator): The educational intervention will be developed with the students, led by the neonatology teacher, in the simulation laboratory. For the training, neonatal high-fidelity simulators, clinical history and paraclinical exams, necessary supplies for the procedure, a simulated mother, a professional nurse and a nursing assistant will be available. Training will take place in individual skill stations (identification of indications, communication, management of medical devices and procedures) and in integrated clinical scenarios.
  Interventions: Other: • Simulated scenario

INTERVENTIONS:
Other: Digital didactic environment — Students assigned to this group will receive access to a digital didactic environment where they will have at their disposal the exchange transfusion guide and a complete video explaining the indications, the preparation of supplies and the newborn for the procedure, the management of medical devices required and a step-by-step description of the exchange transfusion technique. Finally, the student will see an integrated clinical case. This video will be developed by the neonatology and paediatric medical education teaching team in the simulation laboratory of the university using neonatal high-fidelity simulators, a simulated mother and the necessary medical equipment and supplies.
  Arms: Digital didactic environment
Other: • Simulated scenario — The educational intervention will be developed with the students, led by the neonatology teacher, in the simulation laboratory. For the training, neonatal high-fidelity simulators, clinical history and paraclinical exams, necessary supplies for the procedure, a simulated mother, a professional nurse and a nursing assistant will be available. Training will take place in individual skill stations (identification of indications, communication, management of medical devices and procedures) and in integrated clinical scenarios.
  Arms: • Simulated scenario

SUMMARY:
Abstract

Background: Exchange transfusion is a highly complex procedure that requires high levels of expertise. Paediatricians trainees do not have adequate training because opportunities to perform this procedure in practice are scarce. This protocol seeks to compare two educational interventions for exchange transfusions that allow the students to develop competencies to perform the technique in an appropriate and safe way.

Methods/design: A randomized parallel single-blind clinical trial with allocation by simple randomization to the educational intervention (simulation or a digital didactic environment). Students from the paediatric specialization who volunteer to participate will be included. A practical evaluation of the procedure will be performed through a simulated scenario using a standardized clinical case. The main outcome is defined as the result of evaluation using the Objective Structured Clinical Examination; superior performance will be defined when the percentage is greater than or equal to 85%, and nonsuperior performance will be defined when the result is less than 84%. The chi-square independence test or the Fisher exact test will be used to evaluate the effect of the interventions. Multivariate analysis will be performed using a non-conditional logistic regression model. Stata 14 ® software will be used.

Discussion: Exchange transfusion is a procedure that requires expertise to achieve adequate outcomes. The inclusion of new educational strategies, such as simulation and digital didactic environments, is seen as a training option that can improve performance in clinical skills, reduce adverse events and increase the level of trust.

ELIGIBILITY:
Inclusion Criteria:

* o Men and women of legal age who are students enrolled in a paediatrics specialization programme at Colombian university medical schools.

  * Students in any year of specialization in paediatrics.

Exclusion Criteria:

* Students who are, as part of their curriculum, in a rotation outside the country.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2022-08-30 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2024-11-30 (Actual)

PRIMARY OUTCOMES:
Overall result of the OSCE evaluation (checklist). | The checklist was applied by a reviewer blinded to the assignment of the type of intervention by reviewing the video, on average 4 week after of the participation of the groups in the scenarios
  The performance score will be the score obtained for the evaluation divided by the maximum possible score of the test and multiplied by 100. A superior performance is defined as a score greater than or equal to 85%, and a nonsuperior performance is defined as a score equal to or less than 84%.

SECONDARY OUTCOMES:
Performance on the OSCE checklist in sub-areas: Clinical History | The checklist was applied by a reviewer blinded to the assignment of the type of intervention by reviewing the video, on average 4 week after of the participation of the groups in the scenarios
  Clinical history and approach to patient risk and indication for exchange transfusion
Performance on the OSCE checklist in sub-areas: assesment | The checklist was applied by a reviewer blinded to the assignment of the type of intervention by reviewing the video, on average 4 week after of the participation of the groups in the scenarios
  Comprehensive assessment of the patient with neonatal jaundice
Performance on the OSCE checklist in sub-areas: exchange transfusion | The checklist was applied by a reviewer blinded to the assignment of the type of intervention by reviewing the video, on average 4 week after of the participation of the groups in the scenarios
  Management of the patient with neonatal jaundice and indication for exchange transfusion

CONTACTS AND LOCATIONS:
Overall Officials: Maria J Maldonado, Pediatrician, Principal Investigator — Universidad de la Sabana
Locations (1):
- Universidad de La Sabana, Chía, Cundinamarca, Colombia

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available

REFERENCES:
- [Derived] Maldonado MJ, Agudelo SI, Suarez JD, Gamboa O. Educational strategy for the development of skills in exchange transfusion: a randomized clinical trial protocol. Trials. 2020 May 7;21(1):387. doi: 10.1186/s13063-020-04312-3. PMID 32381105